CLINICAL TRIAL: NCT02418390
Title: The Efficacy and Safety of Prophylactic Central Lymph Node Dissection in Papillary Thyroid Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kyu Eun Lee, Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-1404-050-571
Record Dates: First submitted 2015-04-07; First posted 2015-04-16 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Thyroid Cancer, Papillary
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No prophylactic central dissection (No Intervention): Patients underwent total thyroidectomy for papillary thyroid carcinoma, without prophylactic central lymph node dissection
- Prophylactic central dissection (Active Comparator): Patients underwent total thyroidectomy for papillary thyroid carcinoma, with prophylactic central lymph node dissection
  Interventions: Procedure: prophylactic central lymph node dissection

INTERVENTIONS:
Procedure: prophylactic central lymph node dissection — dissection of level VI compartment by AAHNS (American association of head and neck surgeons) classification
  Arms: Prophylactic central dissection

SUMMARY:
The aim of this study is to investigate the efficacy and safety of prophylactic central lymph node dissection in papillary thyroid carcinoma.

DETAILED DESCRIPTION:
The aim of this study is to investigate the efficacy and safety of prophylactic central lymph node dissection in papillary thyroid carcinoma. Primary outcome is the surgical completeness, recurrence rate, and successful ablation rate. Secondary outcomes are the incidence of postoperative complications and PTC stage. The enrolled patients were randomly assigned to control group and intervention group (1:1 allocation).

ELIGIBILITY:
Inclusion criteria were as follows:

1. patients aged 20 to 70 years old
2. patients diagnosed with PTC or suspicious for PTC on fine needle aspiration or core needle biopsy
3. patients with no evidence of LNM before and during surgery(cN0)
4. patients with no evidence of distant metastasis(cM0).

Exclusion criteria were as follows:

1. patients suspected of advanced PTC(clinically T3 or T4) such as invasion of peripheral organs on preoperative examination
2. patients who have previous history of cervical radiation therapy or surgery.
3. pregnant women
4. uncontrolled diabetes, hypertension, or chronic renal failure
5. aspirin or anticoagulant medication within 7 days
6. other clinical trial participation within 30 days
7. radiation exposure to the head and neck
8. previous operation to the neck
9. advanced thyroid cancer including adjacent organ invasion

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2020-10-08 (Actual)

PRIMARY OUTCOMES:
The number of participants with successful surgical completeness | Participants will be followed from the operation to 5 year (maximum)
  In the case of patients undergoing RAI ablation, surgical completeness was defined as cases with a negative ultrasonographic finding with postoperative 1st stimulated Tg <1 ng/mL.
  In patients who did not undergo RAI treatment, the case with a negative finding at the 1st postoperative ultrasound with postoperative 1st unstimulated Tg <0.2ng/mL was defined as surgical completeness.
Recurrence rate of thyroid cancer | Participants will be followed from the operation to 5 year (maximum)
  Recurrence was defined according to the definition of response to therapy in the 2015 American Thyroid Association(ATA) guidelines.
Number of participants with successful ablation | Participants will be followed from the operation to 5 year (maximum)
  Successful ablation was defined as a patient whose stimulated Tg level was measured as <1 ng/mL at last ablation.

SECONDARY OUTCOMES:
postoperative complication occurrence rate | Participants will be followed from the operation to 5 year (maximum)
  At outpatient clinic (6months posteoperatively), video laryngoscopic exam and serum parathyroid hormone with serum calcium will be measured. Type and number of complications will be recorded
impact of prophylactic central lymph node dissection on staging of papillary thyroid cancer(PTC) | TNM stage of each case was confirmed after final pathologic reports. At our facility, final pathologic reports would be turned out at an average of 2 weeks after surgery
  Postoperative complications was divided into transient complication (< 6 months) and permanent complication (≥ 6 months) according to the duration.
  Hypoparathyroidism was diagnosed when patients were given oral calcium supplements to relieve symptoms of hypocalcemia or when serum parathyroid hormone (PTH) levels were lower than baseline values;1) PTH <10 pg/mL on days 1 and 14 after surgery; and 2) PTH <15 pg/mL at least 3 months after surgery.
  All patients underwent a laryngeal ultrasound or laryngoscope after surgery to check for RLN injury. RLN injury was diagnosed when the vocal cord movement was hypomobile or fixed on evaluation. In addition, present study evaluated symptoms related to voice changes, such as hoarseness, thickened voice, difficulty in making high pitch sound, easy voice fatigue, aspiration, or dyspnea in an outpatient clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Kyu Eun Lee, MD, PhD, Principal Investigator — Seoul National University College of Medicine
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carling T, Carty SE, Ciarleglio MM, Cooper DS, Doherty GM, Kim LT, Kloos RT, Mazzaferri EL Sr, Peduzzi PN, Roman SA, Sippel RS, Sosa JA, Stack BC Jr, Steward DL, Tufano RP, Tuttle RM, Udelsman R; American Thyroid Association Surgical Affairs Committee. American Thyroid Association design and feasibility of a prospective randomized controlled trial of prophylactic central lymph node dissection for papillary thyroid carcinoma. Thyroid. 2012 Mar;22(3):237-44. doi: 10.1089/thy.2011.0317. Epub 2012 Feb 7. PMID 22313454